CLINICAL TRIAL: NCT06299098
Title: A Randomized, Double-Blind Study of The Efficacy and Safety of Trevogrumab, With or Without Garetosmab, in Addition to Semaglutide in Patients With Obesity
Brief Title: A Study to Test if Trevogrumab or Trevogrumab With Garetosmab When Taken With Semaglutide is Safe and How Well They Work in Adult Patients With Obesity for Weight Loss, Fat Loss, and Lean Mass Preservation
Acronym: COURAGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1033-OB-2288
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: Obesity without diabetes; Quality of weight loss; Fat mass loss; Lean mass loss
MeSH Terms: conditions — Obesity | interventions — activin A; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Placebo (Placebo Comparator): Part A Randomized 1:1
  Interventions: Drug: Matching Placebo-Part A
- Trevogrumab (Experimental): Part A Randomized 1:1
  Interventions: Drug: Trevogrumab-Part A
- Arm A0 (Experimental): Part B Semaglutide (sema) and subcutaneous (SC) placebo and intravenous (IV) placebo followed by SC placebo Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Semaglutide; Drug: Matching Placebo-Trevogrumab; Drug: Matching Placebo-Garetosmab
- Arm A1 (Experimental): Part B Sema and SC placebo and IV placebo followed by high dose trevogrumab (trevo) Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Semaglutide; Drug: Matching Placebo-Trevogrumab; Drug: Matching Placebo-Garetosmab
- Arm B0 (Experimental): Part B Sema, moderate-high dose trevo, and IV placebo followed by SC placebo Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Semaglutide; Drug: Matching Placebo-Trevogrumab; Drug: Matching Placebo-Garetosmab
- Arm B1 (Experimental): Part B Sema, moderate-high dose trevo, and IV placebo followed by high dose trevo Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Semaglutide; Drug: Matching Placebo-Garetosmab
- Arm C0 (Experimental): Part B Sema, high dose trevo, and IV placebo followed by SC placebo Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Semaglutide; Drug: Matching Placebo-Trevogrumab; Drug: Matching Placebo-Garetosmab
- Arm C1 (Experimental): Part B Sema, high dose trevo, and IV placebo followed by high dose trevo Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Semaglutide; Drug: Matching Placebo-Garetosmab
- Arm D0 (Experimental): Part B Sema, high dose trevo, and garetosmab (gareto) followed by SC placebo Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Garetosmab; Drug: Semaglutide; Drug: Matching Placebo-Trevogrumab
- Arm D1 (Experimental): Part B Sema, high dose trevo, and gareto followed by high dose trevo Randomized 1:1:1:1:1:1:1:1
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Garetosmab; Drug: Semaglutide
- Arm 1 (Experimental): Part C Sema and SC placebo Randomized 1:2:2
  Interventions: Drug: Semaglutide; Drug: Matching Placebo-Trevogrumab
- Arm 2 (Experimental): Part C Sema and SC low dose trevo Randomized 1:2:2
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Semaglutide; Drug: Matching Placebo-Trevogrumab
- Arm 3 (Experimental): Part C Sema and SC moderate dose trevo Randomized 1:2:2
  Interventions: Drug: Trevogrumab-Part B and Part C; Drug: Semaglutide

INTERVENTIONS:
Drug: Trevogrumab-Part A — Administered IV or SC in Part A
  Other Names: REGN1033; GDF8
  Arms: Trevogrumab
Drug: Trevogrumab-Part B and Part C — Administered SC in Part B, Part C
  Other Names: REGN1033; GDF8
  Arms: Arm 2; Arm 3; Arm A1; Arm B0; Arm B1; Arm C0; Arm C1; Arm D0; Arm D1
Drug: Garetosmab — Administered IV in Part B
  Other Names: REGN2477; Activin A
  Arms: Arm D0; Arm D1
Drug: Semaglutide — Administered SC in Part B and Part C
  Other Names: Wegovy®
  Arms: Arm 1; Arm 2; Arm 3; Arm A0; Arm A1; Arm B0; Arm B1; Arm C0; Arm C1; Arm D0; Arm D1
Drug: Matching Placebo-Part A — Administered IV or SC in Part A
  Arms: Placebo
Drug: Matching Placebo-Trevogrumab — Administered SC in Part B and Part C
  Arms: Arm 1; Arm 2; Arm A0; Arm A1; Arm B0; Arm C0; Arm D0
Drug: Matching Placebo-Garetosmab — Administered IV in Part B
  Arms: Arm A0; Arm A1; Arm B0; Arm B1; Arm C0; Arm C1

SUMMARY:
This study is researching experimental drugs called trevogrumab and garetosmab (called "study drugs") in combination with another drug, semaglutide (Wegovy®). This study will be done in 3 parts, Part A, Part B, and Part C where different study drugs will be tested.

Part A of the study is focused on healthy participants. Part B and C of the study is focused on participants with obesity.

The aim of Part A of the study is to see how safe and tolerable the study drug is in healthy participants. The aim of Part B and Part C of the study is to see how safe and effective the study drug is when combined with Wegovy.

Parts A, B, and C of the study are looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

DETAILED DESCRIPTION:
Part A Healthy Volunteers

Part B and Part C (starts after treatment for Part A has completed) Participants with Obesity

ELIGIBILITY:
Key Inclusion Criteria

Part A

1. Male or female participants age ≥18 to ≤55 years of age at the time of screening
2. BMI ≥18 and ≤32 kg/m2, at the screening visit

   Part B and Part C
3. Male or female participants ≥18 to ≤80 years of age at the time of screening
4. BMI ≥30 kg/m2, at the screening visit
5. History of 1 or more self-reported unsuccessful dietary attempts to lose weight

Key Exclusion Criteria

1. History of diabetes (Type 2 or Type 1). History of gestational diabetes is permitted
2. Previous bariatric surgery or planned bariatric surgery
3. History of hypertrophic cardiomyopathy
4. Abnormal electrocardiogram (ECG) findings at screening that meet Cornell voltage criteria for left ventricular hypertrophy
5. Any malignancy in the past 5 years prior to screening (except for nonmelanoma skin cancer that has been resected with no evidence of metastatic disease for 3 years prior to screening)
6. History of poorly controlled hypertension, as defined in the protocol
7. Have a history of any other condition (such as known drug abuse, alcohol abuse, diagnosed eating disorder, or a severe mental illness) that, in the opinion of the investigator, may preclude the participant from following and completing the protocol
8. Have history of use of marijuana/tetrahydrocannabinol (THC) within 90 days prior to Visit 1 of enrollment and are unwilling to abstain from marijuana/THC use during the trial
9. Has a history of any neuromuscular disorder (eg, multiple sclerosis, myasthenia gravis, myopathy, peripheral neuropathy, etc)

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to week 7
  Part A
Severity of TEAEs | Baseline to week 7
  Part A
Percent change in total fat mass | Baseline to week 26
  Part B
Percent change in total lean mass | Baseline to week 26
  Part B
Percent change in body weight | Baseline to week 26
  Part B
Percent change in total fat mass | Baseline to week 52
  Part C
Percent change in total lean mass | Baseline to week 52
  Part C
Percent change in body weight | Baseline to week 52
  Part C

SECONDARY OUTCOMES:
Concentrations of trevogrumab in serum over time | Up to 75 weeks
  Part A, Part B, and Part C
Percent change in total fat mass | Baseline to week 52
  Part B
Percent change in total lean mass | Baseline to week 52
  Part B
Percent change in body weight | Baseline to week 52
  Part B
Change in waist circumference (cm) | Baseline to week 26
  Part B and Part C
Change in waist circumference (cm) | Baseline to week 52
  Part C
Percent change in fasting serum triglycerides | Baseline to week 26
  Part B
Percent change in total cholesterol | Baseline to week 26
  Part B
Percent change in Apolipoprotein B (Apo B) | Baseline to week 26
  Part B
Percent change in Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline to week 26
  Part B
Concentrations of garetosmab in serum over time | Up to 75 weeks
  Part B
Incidence of anti-drug antibodies (ADA) to trevogrumab after repeated doses over time | Up to 75 weeks
  Part B and Part C
Magnitude of ADAs to trevogrumab over time | Up to 75 weeks
  Part B and Part C
Incidence of ADAs to garetosmab after repeated doses over time | Up to 75 weeks
  Part B
Magnitude of ADAs to garetosmab over time | Up to 75 weeks
  Part B
Incidence of TEAEs | Up to 75 weeks
  Part B and Part C
Severity of TEAEs | Up to 75 weeks
  Part B and Part C
Percent change in total fat mass | Baseline to week 26
  Part C
Percent change in total lean mass | Baseline to week 26
  Part C
Percent change in body weight | Baseline to week 26
  Part C
Concentration of total Growth Differentiation Factor (GDF) 8 in serum over time | Up to 75 weeks
  Part C

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (60):
- United States (58):
  - Pinnacle Research Group, Anniston, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Foothills Research Center Cct Research, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - ProSciento, Chula Vista, California
  - Valiance Clinical Research- Huntington Park, Huntington Park, California
  - Velocity, San Diego, La Mesa, California
  - Northern California Research, Sacramento, California
  - Acclaim Clinical Research, San Diego, California
  - Metabolic Institute of America, Tarzana, California
  - Valiance Clinical Research, Tarzana, California
  - Southwest General Healthcare Center, Fort Myers, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - IMA Clinical Research St. Petersburg, St. Petersburg, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Clinical Research of Central Florida - Bond Clinic, Winter Haven, Florida
  - Center for Advanced Research and Education, Gainesville, Georgia
  - Balanced Life Health Care Solutions, Lawrenceville, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Prairie Education and Research Cooperative (PERC), Springfield, Illinois
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - IMA Clinical Research Monroe - Armand, Monroe, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Prime Health and Wellness Clinic, Fayette, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Sky Integrative Medical Center Skycrng, Ridgeland, Mississippi
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Clinvest Research, Springfield, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Hassman Research Institute, Berlin, New Jersey
  - Accellacare Clinical Research, Raleigh Medical Group, Raleigh, North Carolina
  - Accellacare of Salisbury, Salisbury, North Carolina
  - Accellacare of Piedmont, Piedmont Healthcare, Statesville, North Carolina
  - Pmg Research of Wilmington Llc, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Javara Incorporated at Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Velocity Clinical Research Inc., Cincinnati, Ohio
  - AMR Norman, Norman, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Tribe Clinical Research Llc, Greenville, South Carolina
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - Pmg Research of Bristol, Bristol, Tennessee
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - PMG Research of Knoxville - Merchant Drive, Knoxville, Tennessee
  - PMG Research of Knoxville - Emory Road, Knoxville, Tennessee
  - Velocity Clinical Research Dallas, Dallas, Texas
  - Medresearch Inc, El Paso, Texas
  - Valley Institute of Research, Fort Worth, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
- Puerto Rico (2):
  - Fundacion de Investigacion (FDI) Clinical Research, San Juan
  - PRCCI Clinical Research Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: Courage Study — https://couragestudy.com/en-us/home/